CLINICAL TRIAL: NCT01777386
Title: Perforator Artery Changes During Suprafascial Pre-expansion of the Perforator Flaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emre Hocaoglu, Dr., Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hocaoglupreexpandedperforator1
Record Dates: First submitted 2013-01-18; First posted 2013-01-28 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Scar; Contracture; Flap Disorder
Keywords: scar; contracture; perforator flap; preexpanded perforator flap; perforator vessel; artery diameter
MeSH Terms: conditions — Cicatrix; Contracture

ARMS (2):
- preexpanded flap (Active Comparator): Fourteen patients were treated with fifteen '' preexpanded perforator flap surgery '' interventions. The last six cases were evaluated in terms of perforator artery diameter before and after expansion process. The preexpanded flap donor sites' perforator artery diameters were also compared with their anatomic equivalents located in the symmetric side of the body.
  Interventions: Procedure: preexpanded perforator flap surgery
- control side (No Intervention): In six of the 14 patients, perforator artery diameter of the nonexpanded symmetric anatomical side of the body (equivalent to the expanded site)were measured.

INTERVENTIONS:
Procedure: preexpanded perforator flap surgery
  Arms: preexpanded flap

SUMMARY:
Tissue expansion methods have been recommended as a means of improving the clinical results with perforator flaps but in plastic surgery literature there are few clinical trials supporting this opinion. The purposes of this clinical study are to address the ''preexpanded perforator flap concept'' by demonstrating a case series of relevant reconstructive procedures and to evaluate the perforator vessel changes that happen during the expansion periods of various perforator flap donor sites.

ELIGIBILITY:
Inclusion Criteria:

* patients with broad scars and contracture bands
* patients with esophagocutaneous fistula
* patients with ambiguous genitalia

Exclusion Criteria:

* none

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Transferred tissue dimensions | At least five months after the operation
  Demonstrating the amount of transferred healthy tissue exhibits the success of the technique.

SECONDARY OUTCOMES:
Diameter of the perforator artery in a particular tissue level | Measured the day before the expander implantation surgery and the day before the flap transfer surgery (second session following tissue expansion)
  This measurement will reveal one of the morphologic changes happen during tissue expansion period (perforator flap preexpansion). This measurement will be done for the last six patients. The diameter of the perforator artery of the preexpanded flap will be compared with both the diameter of the same artery before the expansion process and the diameter of the equivalent perforator artery of the symmetric side (non expanded side)of the body.